CLINICAL TRIAL: NCT03824470
Title: The Effect of Non-Muscle Intubation on Post Operative Recovery Conditions in Patients With Obstructive Sleep Apnea Syndrome: Double Blind Randomized Controlled Study
Brief Title: The Effect of Intubation Without Muscle Relaxation on Post Operative Recovery Conditions: Double Blind Randomized Controlled Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Celaleddin Soyalp, Assist. prof., Yuzuncu Yil University
Other Study IDs: stop bang
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: stop bang; Intubation Without Muscle Relaxation; Post Operative Recovery; TOF
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group E(rocuronium): E, after the administration of 1 mg / kg lidocaine, 2 mg / kg propofol, 1 mcg / kg remifentanil and 0.6 mg / kg rocuronium intravenously, patients will be intubated and general anesthesia will be performed when the Tof value is 0.
- Group R (remifentanil): 1 mg / kg lidocaine, 4 mcg / kg remifentanil and 2 mg / kg propofol intravenously.patients will be intubated and general anesthesia will be performed when the Tof value is 0

SUMMARY:
The primary aim of this study is to research the effect of intubation without muscle relaxant on post-operative recovery conditions in patients with OSAS (obstructive sleep apnea syndrome). Our secondary aim is to research the hemodynamic parameters in intraoperative period and complications such as sore throat and laryngospasm voice limitation in the postoperative period.

DETAILED DESCRIPTION:
Study Protocol, Methods and Procedures to be Applied:

This study will be carried out as double blinded randomized controlled after the approval of the ethics committee of our hospital. By carrying out the Stop Bang questionnaire which is a practical and highly sensitive test, 60 patients ranging from 18 to 65 years with a stop bang score of 3 and ASA I-II and mallampati I and II scores will be included to the study. The patients included in the study will be divided into two groups of 30 people randomly with a closed envelope method. Patients who were intubated in the intensive care unit during postoperative period, those using CPAP device at home or those who received OSAS therapy, who had undergone head and neck surgery or who had head surgery, central nervous system damage and cardiovascular or pulmonary stability, neuromuscular disease patients, those with known allergies to the anesthetic agents used, those whose written and verbal consent cannot be obtained, smokers, pregnants and patients with ASA III and IV will not be included in our study. All patients will be seen a day in advance and after performing stop bang test, those with test score of 3 and above will be included in the study and their physical examinations and laboratory findings will be evaluated. The demographic data of the patients will be recorded. The physician performing the anesthesia and the evaluating physician will be different people. The evaluating physician will not know which anesthetic agent is used to the patients. The group to be performed Esmeron will be named Group E and the group to be given Remifentanil will be named Group R. All patients included in the study will be taken to the operation room and the hemodynamic parameters (heart rate, mean blood pressure values, SpO2) will be recorded by naninvasive monitoring. The data obtained will be considered as basal. All patients will be given 2 mg / kg demisolam for the purpose of sedation. General anesthesia will be done by connecting the Tof device to the patients. Anesthesia induction will be done to anesthesia induction Group R with 1 mg / kg lidocaine, 4 mcg / kg remifentanil and 2 mg / kg propofol intravenously. In group E, after the administration of 1 mg / kg lidocaine, 2 mg / kg propofol, 1 mcg / kg remifentanil and 0.6 mg / kg rocuronium, patients in both groups will be intubated and general anesthesia will be performed when the Tof value is 0. During intubation; intubation difficulty will be evaluated and recorded by intubation scoring system. Anesthesia maintenance in both groups will be provided with 8% desflurane, 40% O2, 60% dry air and iv. 0.025 mcg / kg / min remifentanil fusion. During the study, the recorded basal hemodynamic parameters of the patients will be recorded in the first 20 minutes of the operation with a 5-minute interval and 10-minute interval after the 20th minute. In case of a change of 20% in any one according to basal, it will be intervened immediately. In order to provide the depth of anesthesia before the operation, patients will be monitored with TOF device and the depth of anesthesia will be provided. Shortly after the end of the surgery, the gases will be cut off and the Tof value of 70% and above will be recorded. When Tof is 70%, Group R will be given 10 cc physiological saline intravenously. In order to antagonize the muscle relaxant effect in Group E, 2 / mg / kg sguamadex will be administered intravenously by diluting with 10 cc physiological saline. Patients will be extubated when the tof value of both groups is 90%. The durations from 70% to 90% of the Tof value, spontaneous eye opening duration after the patient is extubated, duration of extubation, response duration to commands, duration until modified aldrete score is 10, surgeon satisfaction (good, bad, moderate) and duration of surgery will be recorded. The operation will be terminated by recording whether there is a need for ventilation with sore throat, laryngospasm volume restriction, desaturation and mask.

ELIGIBILITY:
Inclusion Criteria:

Aged18- 65 years With a stop bang score of 3 ASA I-II Mallampati I and II scores

Exclusion Criteria:

* Patients who were intubated in the intensive care unit during postoperative period, those using CPAP device at home or those who received OSAS therapy, who had undergone head and neck surgery or who had head surgery, central nervous system damage and cardiovascular or pulmonary stability, neuromuscular disease patients, those with known allergies to the anesthetic agents used, those whose written and verbal consent cannot be obtained, smokers, pregnants and patients with ASA III and IV will not be included in our study.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: the patiens whose Stop Bang questionnaire bigger tan 3 and planned for elective surgery
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-02-05 (Estimated); Primary Completion 2019-03-15 (Estimated); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
Post Operative Recovery | 1 hour
  The durations from 70% to 90% of the Tof value, spontaneous eye opening duration after the patient is extubated, duration of extubation, response duration to commands, duration until modified aldrete score is 10

CONTACTS AND LOCATIONS:
Overall Officials: CELALEDDİN Y SOYALP, Study Chair — Yuzuncu Yil University

IPD SHARING:
Plan to Share IPD: Undecided